CLINICAL TRIAL: NCT06957834
Title: Randomised Double-blinded Split-face Controlled Study to Evaluate the Effectiveness of Eflornithine Hydrochloride Cream Compared to Topical Hydroquinone 2% Cream for the Treatment of Melasma.
Brief Title: Efficacy of Eflornithine Hydrochloride Cream in the Treatment of Melasma: A Randomized, Double-blinded, Split-face Controlled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Skin Centre (Network)
Responsible Party: Principal Investigator, Steven Thng Tien Guan, Deputy Director and Senior Consultant, National Skin Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/00399
Record Dates: First submitted 2025-05-02; First posted 2025-05-05 (Actual); Last update posted 2025-05-05 (Actual); Status verified 2025-05

CONDITIONS: Melasma
Keywords: Melasma; Dermatology; Eflornithine
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, split-face study. Both treatments (Eflornithine hydrochloride, and Hydroquinone) will be applied simultaneously: one on the left side of the face and the other on the right side. Treatment allocation to facial sides will be randomized, and participants blinded (both treatments with similar packaging, look and consistency). Outcomes will be assessed on each side of the face by a blinded evaluator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eflornithine hydrochloride cream on right half of face, Hydroquinone cream on left half of face (Active Comparator)
  Interventions: Drug: Eflornithine hydrochloride cream; Drug: Hydroquinone cream
- Eflornithine hydrochloride cream on left half of face, Hydroquinone cream on right half of face (Active Comparator)
  Interventions: Drug: Eflornithine hydrochloride cream; Drug: Hydroquinone cream

INTERVENTIONS:
Drug: Eflornithine hydrochloride cream — Eflornithine hydrochloride cream at 11.5% applied twice daily
Drug: Hydroquinone cream — Hydroquinone 2% cream, applied twice daily

SUMMARY:
The goal of this clinical trial is to learn if Eflornithine hydrochloride cream works to treat melasma in adults, in comparison to Hydroquinone cream. It will also learn about the safety of Eflornithine hydrochloride cream. The main questions it aims to answer are:

* Does Eflornithine hydrochloride improve melasma assessment scores over a 3-month duration compared to Hydroquinone cream?
* What side effects might patients get while using Eflornithine hydrochloride cream?

Participants will:

* Apply both Eflornithine hydrochloride and Hydroquinone creams on separate halves of their faces every day for 3 months.
* Visit the clinic once at the 2-month mark and once at the 3-month mark for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of melasma
* Fitzpatrick Type III or IV
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or lactating patients
* Patients with difficulty adhering to regular topical treatments
* Patients with known contact allergies to any of the ingredients in the topical medications used in the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Modified Melasma Area and Severity Index (mMASI) | At 8 weeks and 12 weeks
Mexameter melanin score | At 8 and 12 weeks
  Mexameter device (Courage + Khazaka Electronic GmbH, Germany)

SECONDARY OUTCOMES:
Mexameter erythema score | At 8 and 12 weeks
  Mexameter device (Courage + Khazaka Electronic GmbH, Germany)
Patient Satisfaction Score | At 8 and 12 weeks
  For each side of the face, each patient and dermatologist was asked to grade the severity of melasma from a score of 0 (cleared), 1 (mild), 2 (moderate) to 3 (severe)
Physician Global Assessment | At 8 and 12 weeks
  For each side of the face, each patient and dermatologist was asked to grade the severity of melasma from a score of 0 (cleared), 1 (mild), 2 (moderate) to 3 (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- National Skin Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in publication
Time Frame: Beginning 6 months and ending 2 years after publication
Access Criteria: Upon reasonable request to corresponding author